CLINICAL TRIAL: NCT03252886
Title: The Efficacy of Videolaryngoscopy During Cardiac-pulmonary Resuscitation (CPR) for Trauma Patients With Suspect Neck Injuries
Brief Title: Videolaryngoscopy During CPR for Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRAUMACPRintu
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cardiopulmonary Arrest; Neck Injury Multiple
Keywords: intubation; Cardiopulmonary Resuscitation; neck injury
MeSH Terms: conditions — Heart Arrest; Neck Injuries | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DL user (Active Comparator): Experienced emergency physicians who primarily use the direct laryngoscopy (DL) for endotracheal intubation during cardio-pulmonary resuscitation.
  Interventions: Procedure: Endotracheal Intubation
- VL user (Active Comparator): Experienced emergency physicians who primarily use the videolaryngoscopy (VL) for endotracheal intubation during cardio-pulmonary resuscitation.
  Interventions: Procedure: Endotracheal Intubation

INTERVENTIONS:
Procedure: Endotracheal Intubation — Insertion of endotracheal tube into the trachea and supply oxygen using the Ambu-bagging during cardiopulmonary resuscitation

SUMMARY:
This is a clinical study based on collected video-clip data of cardiopulmonary resuscitation for patients with suspected neck injury in multiple trauma between 2011 and 2015. The study aimed to compare all possible factors relating to ETI performance during CPR for truma patients between experienced video-laryngoscopy and direct- laryngoscopy users.

DETAILED DESCRIPTION:
Endotracheal intubation (ETI) is considered to be the best method of airway management during cardiopulmonary resuscitation (CPR). However ETI during CPR is a highly skill-dependent procedure, then it should be attempted only highly trained physicians. Especially, cervical immobilization by neck collar in truamatic patients is a great obstacle to successful ETI during CPR.

Because of technical difficulty in using direct laryngoscopy (DL), various types of videolaryngoscopy (VL) devices have been developed to overcome the problems of DL. VL may be more useful to perform ETI during CPR for trauma patients with cervical immobilization.

This study tried to compare the success rate of endotracheal intubation (ETI), speed of ETI, incidence of complications, and chest compression interruptions during cardiopulmonary resuscitation for trauma patients with suspected neck injury between intubators using the DL and the VL in a real clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Multiple trauma patients with suspected neck injuries
* Arrest Patients

Exclusion Criteria:

* Case of requesting the do-not attempt resuscitation before ETI
* already intubated case before arrival to hospital
* Cardiac arrest from non-traumatic causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
First attempt successful ETI | within 1 hour after emergency department visit
  Successfully insertion of endotracheal tube into trachea at first attempt

SECONDARY OUTCOMES:
the time to complete ETI from the beginning | within 1 hour after emergency department visit
  the time from the advancement of the blade into the patient's mouth to the delivery of the first successful ventilation using the bag
Occurance of complication | within 1 hour after emergency department visit
  Presence of chest compression interruption, esophageal intubation and dental injuries

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, M.D,Ph.D, Principal Investigator — School of Medicine, Konkuk University
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea